CLINICAL TRIAL: NCT03038022
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Placebo Controlled Study of MGL-3196 in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Study of MGL-3196 in Patients With Heterozygous Familial Hypercholesterolemia (HeFH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGL-3196-06; 2016-002315-17 (EudraCT Number)
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Heterozygous Familial Hypercholesterolemia
MeSH Terms: interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MGL-3196 (Experimental): Study Drug
  Interventions: Drug: MGL-3196 (resmetirom)
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MGL-3196 (resmetirom) — Oral
  Arms: MGL-3196
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of once-daily oral MGL-3196 on the percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in participants with Heterozygous Familial Hypercholesterolemia (HeFH).

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate in the study and provide written informed consent;
* Male and female adults ≥18 years of age;
* Female participants of child bearing potential with negative serum pregnancy (beta human chorionic gonadotropin) test who are not breastfeeding, do not plan to become pregnant during the study, and agree to use effective birth control per locally agreed requirements; male participants who have sexual intercourse with a female partner of child bearing potential from the first dose of study drug until 1 month after study completion must either be surgically sterile (confirmed by documented azoospermia >90 days after the procedure) or agree to use a condom with spermicide. All male participants must agree not to donate sperm from the first dose of study drug until 1 month after study completion;
* Must have a diagnosis of HeFH by genetic testing or by having met the diagnostic criteria for definite familial hypercholesterolemia outlined by the Simon Broome Register Group or World Health Organization/Dutch Lipid Network (score >8);
* Must have had a fasting LDL-C (low density lipoprotein cholesterol) ≥2.6 mmol/L (100 mg/dL); and
* Must be on a stable or maximally tolerated dose (≥4 weeks prior to screening) of an approved statin (rosuvastatin ≤40 mg daily, atorvastatin ≤80 mg daily), with or without ezetimibe. Patients intolerant to statins were allowed.

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* LDL or plasma apheresis within 2 months prior to randomization;
* New York Heart Association class III or IV heart failure, or known left ventricular ejection fraction <30%;
* Uncontrolled cardiac arrhythmia, including confirmed QT interval corrected using Fridericia's formula >450 msec for males and >470 msec for females at the screening electrocardiogram assessment;
* Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, or stroke within 3 months prior to randomization;
* Type 1 diabetes, or newly diagnosed or uncontrolled type 2 diabetes (hemoglobin A1c >8%);
* History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening; Note: Significant alcohol consumption is defined as average of >20 g/day in female participants and >30 g/day in male participants;
* Hyperthyroidism;
* Thyroid replacement therapy;
* Hypothyroidism;
* Evidence of chronic liver disease;
* Hepatitis B, as defined by the presence of hepatitis B surface antigen;
* Hepatitis C, as defined by the presence of hepatitis C virus (HCV) antibody (anti-HCV) and HCV ribonucleic acid (RNA). Participants with positive anti-HCV who test negative for HCV RNA at screening will be allowed to participate in the study;
* Serum alanine aminotransferase >1.5 x upper limit of normal (ULN) (one repeat allowed);
* Estimated glomerular filtration rate <60 mL/min;
* Creatine kinase >3 x ULN (one repeat allowed);
* History of biliary diversion;
* Positive for human immunodeficiency virus infection;
* History of malignant hypertension;
* Systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg at screening or randomization and confirmed at an unscheduled visit;
* Triglycerides >5.7 mmol/L (500 mg/dL) at screening and confirmed by repeat assessment;
* Active, serious medical disease with likely life expectancy <2 years;
* Active substance abuse, including inhaled or injection drugs within the year prior to screening;
* Participation in an investigational new drug trial within the 30 days prior to randomization; or
* Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, or compromise the well-being of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — Madrigal Pharmaceuticals, Inc.
Locations (13):
- Denmark (5):
  - Madrigal Research Site, Aalborg
  - Madrigal Research Site, Copenhagen
  - Madrigal Research Site, Esbjerg
  - Madrigal Research Site, Herlev
  - Madrigal Research Site, Viborg
- Netherlands (6):
  - Madrigal Research Site, Amsterdam
  - Madrigal Research Site, Apeldoorn
  - Madrigal Research Site, Goes
  - Madrigal Research Site, Hoorn
  - Madrigal Research Site, Nijmegen
  - Madrigal Research Site, Zwijndrecht
- Norway (2):
  - Madrigal Research Site - 1, Oslo
  - Madrigal Research Site - 2, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovingh GK, Klausen IC, Heggen E, McCarty K, Zhou R, Isaac BF, Taub R, Langslet G, Kastelein JJP. Resmetirom (MGL-3196) in Patients With Heterozygous Familial Hypercholesterolemia. J Am Coll Cardiol. 2022 Mar 29;79(12):1220-1222. doi: 10.1016/j.jacc.2022.01.023. No abstract available. PMID 35331419

RESULTS

PARTICIPANT FLOW:
Groups:
- MGL-3196: Participants randomized to MGL-3196 received 100 mg daily during the first 2 weeks, 60 mg daily during Weeks 2 to 4, and then either 60 or 100 mg daily to Week 12 based on Week 2 measured pharmacokinetic (PK) assessments of MGL-3196 exposure.
- Placebo: Participants administered matching oral placebo once daily for 12 weeks.
Period: Overall Study
Arm/Group | MGL-3196 | Placebo
Started | 78 | 38
Received at Least 1 Dose of Study Drug | 78 | 38
Completed | 72 | 36
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- MGL-3196: Participants randomized to MGL-3196 received 100 mg daily during the first 2 weeks, 60 mg daily during Weeks 2 to 4, and then either 60 or 100 mg daily to Week 12 based on Week 2 measured PK assessments of MGL-3196 exposure.
- Total: Total of all reporting groups
Arm/Group | MGL-3196 | Placebo | Total
Number analyzed (Participants) | 78 | 38 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 25 | 81
  >=65 years | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (12.38) | 59.1 (11.33) | 57.3 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 16 | 55
  Male | 39 | 22 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 78 | 38 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 78 | 37 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Low-density Lipoprotein Cholesterol (LDL-C) (Direct measure or ultracentrifugation) [Mean (Standard Deviation); unit: mg/dL] | 131.4 (47.24) | 137.0 (57.53) | 133.3 (50.65)
Statin Use [Count of Participants; unit: Participants]
  Atorvastatin | 40 | 16 | 56
  Rosuvastatin | 34 | 17 | 51
  Pravastatin | 1 | 1 | 2
  None | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in LDL-C From Baseline To Week 12
Description: LDL-C was determined by ultracentrifugation or direct measure. Least-squares (LS) mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Population: Modified Intent-to-Treat (mITT) population: all participants who were randomized in the study, received at least 2 weeks of study drug, and had a valid lipid measurement at Week 2 or later.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -10.6 (2.59) | 8.2 (3.71)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in LDL-C between MGL-3196 and placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -18.8, 95% CI 2-sided [-27.8 to -9.8], Standard Error of Mean 4.52

2. Secondary Outcome: Mean Change From Baseline to Week 12 of Free Thyroxine (T4)
Description: T4 was assessed at each study visit.
Time Frame: Baseline up to Week 12
Population: Safety population: all participants who were randomized in the study and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
ng/dL | -0.268 (0.0130) | 0.009 (0.0185)

3. Secondary Outcome: Mean Change From Baseline to Week 12 of Free Triiodothyronine (T3)
Description: Free T3 was assessed at each study visit.
Time Frame: Baseline up to Week 12
Population: Safety population: all participants who were randomized in the study and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
ng/L | -0.04 (0.038) | 0.10 (0.054)

4. Secondary Outcome: Mean Change From Baseline to Week 12 of Thyrotropin (TSH)
Description: TSH was assessed at each study visit.
Time Frame: Baseline up to Week 12
Population: Safety population: all participants who were randomized in the study and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mIU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
mIU/L | -0.027 (0.0690) | 0.114 (0.0987)

5. Secondary Outcome: Mean Change From Baseline to Week 12 of Thyroxine Binding Globulin (TBG)
Description: TBG was assessed at all study visits except the Screening Visit.
Time Frame: Baseline up to Week 12
Population: Safety population: all participants who were randomized in the study and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
mg/L | -2.31 (0.256) | -0.44 (0.367)

6. Secondary Outcome: Mean Change From Baseline to Week 12 of Reverse Triiodothyronine (T3)
Description: Reverse T3 was assessed at each study visit.
Time Frame: Baseline up to Week 12
Population: Safety population: all participants who were randomized in the study and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
ng/dL | -4.36 (0.392) | -0.58 (0.554)

7. Secondary Outcome: Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 12
Description: Non-HDL-C were determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -12.0 (2.41) | 7.5 (3.46)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -19.5, 95% CI 2-sided [-27.9 to -11.1], Standard Error of Mean 4.22

8. Secondary Outcome: Mean Percent Change In Triglycerides From Baseline To Week 12
Description: Triglycerides were determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Population: mITT population: all participants who were randomized in the study, received at least 2 weeks of study drug, and had a valid lipid measurement at Week 2 or later.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -18.3 (3.24) | 7.2 (4.64)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in triglycerides between MGL-3196 and placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -25.4, 95% CI 2-sided [-36.7 to -14.2], Standard Error of Mean 5.66

9. Secondary Outcome: Mean Percent Change In Lipoprotein(a) (Lp[a]) From Baseline To Week 12
Description: Lp(a) was determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -21.8 (2.87) | 4.4 (4.11)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in Lp(a) between MGL-3196 and placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -26.3, 95% CI 2-sided [-36.2 to -16.4], Standard Error of Mean 5.01

10. Secondary Outcome: Mean Percent Change in Apolipoprotein CIII From Baseline to Week 12
Description: Apolipoprotein CIII was determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -19.3 (2.9) | 3.4 (4.1)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -22.7, 95% CI 2-sided [-32.6 to -12.8]

11. Secondary Outcome: Mean Percent Change In Apolipoprotein B (ApoB) From Baseline To Week 12
Description: ApoB was determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -14.2 (1.66) | 3.8 (2.37)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in ApoB between MGL-3196 and placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -18.0, 95% CI 2-sided [-23.7 to -12.2], Standard Error of Mean 2.90

12. Secondary Outcome: Mean Percent Change in Apolipoprotein B/Apolipoprotein A1 (ApoB/ApoA1) Ratio From Baseline to Week 12
Description: The ApoB/ApoA1 ratio was determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -5.0 (1.8) | 4.2 (2.5)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.0037, ANOVA; Mean Difference (Net) = -9.1, 95% CI 2-sided [-15.3 to -3.0]

13. Secondary Outcome: Mean Percent Change In Cholesterol/HDL-C Ratio From Baseline to Week 12
Description: The Cholesterol/HDL-C Ratio was determined by ultracentrifugation. LS mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change | -3.5 (2.3) | 6.3 (3.3)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.017, ANOVA; Mean Difference (Net) = -9.8, 95% CI 2-sided [-17.8 to -1.8]

14. Secondary Outcome: Absolute Change in LDL-C From Baseline to Week 12
Description: LDL-C was determined by ultracentrifugation or direct measure . Least-squares (LS) mean was provided for the comparison of MGL-3196 versus placebo and it used a linear model with percent change from baseline as the dependent variable and treatment as a factor.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
mg/dL | -17.0 (3.31) | 9.9 (4.74)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -27.0, 95% CI 2-sided [-38.4 to -15.5], Standard Error of Mean 5.79

15. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 2 and Week 4 in Patients in the 100 mg and the 60 mg Groups
Description: as for outcome 1
Time Frame: Baseline to Week 2 and Week 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 76 | 37
percent change
  Week 2 | -16.6 [-22.6 to -10.6] | 1.6 [-3.2 to 6.5]
  Week 4 | -9.8 [-16.3 to -3.4] | 0.1 [-5.2 to 5.4]

16. Secondary Outcome: Percent Change in LDL-C From Baseline to Week 12 by Systemic Exposure Category
Description: The effect on percent change in LDL-C from baseline to Week 12 was determined by patient exposure category (higher/lower). Patients taking MGL-3196 were categorized into lower and higher exposure groups. Patients in the higher exposure group must either have had estimated Week 2 AUC ≥5,000 mg∙h/L, or if Week 2 AUC <5,000 mg∙h/L but Week 4 pre-dose concentration >1.5 ng/mL (if on 60 mg MGL-3196). All other patients were in the lower exposure group.
Time Frame: Baseline to Week 12
Population: mITT Population
Measure: Mean (Standard Error); unit: percent change
Groups:
- MGL-3196 Lower Exposure: Participants randomized to MGL-3196 received 100 mg daily during the first 2 weeks, 60 mg daily during Weeks 2 to 4, and then either 60 or 100 mg daily to Week 12 based on Week 2 measured pharmacokinetic (PK) assessments of MGL-3196 exposure.
- MGL-3196 Higher Exposure: Participants randomized to MGL-3196 received 100 mg daily during the first 2 weeks, 60 mg daily during Weeks 2 to 4, and then either 60 or 100 mg daily to Week 12 based on Week 2 measured pharmacokinetic (PK) assessments of MGL-3196 exposure.
  Patients in the higher exposure group must either have had estimated Week 2 AUC ≥5,000 mg∙h/L, or if Week 2 AUC <5,000 mg∙h/L but Week 4 pre-dose concentration >1.5 ng/mL (if on 60 mg MGL-3196)
Arm/Group | MGL-3196 Lower Exposure | MGL-3196 Higher Exposure | Placebo
Number analyzed (Participants) | 37 | 39 | 37
percent change | -8.1 (3.71) | -13.0 (3.62) | 8.2 (3.71)
Statistical Analysis 1: Comparison: MGL-3196 Lower Exposure vs Placebo; Test type: Superiority; p = 0.0025, ANOVA; Mean Difference (Net) = -16.3, 95% CI 2-sided [-26.7 to -5.9], Standard Error of Mean 5.25
Statistical Analysis 2: Comparison: MGL-3196 Higher Exposure vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -21.2, 95% CI 2-sided [-31.4 to -10.9], Standard Error of Mean 5.18

17. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: Total LDL Particles
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for LDL Particles.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nmol/L | 1223 (334) | 1428 (475)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -245.2, 95% CI 2-sided [-363.7 to -126.7]

18. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: Small LDL Particles
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for Small LDL Particles.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nmol/L | 655 (214) | 760 (265)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.0067, ANOVA; Mean Difference (Net) = -99.4, 95% CI 2-sided [-170.6 to -28.2]

19. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: Intermediate LDL Particles
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for Intermediate LDL Particles.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nmol/L | 157 (96) | 168 (184)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.5245, ANOVA; Mean Difference (Net) = -14.7, 95% CI 2-sided [-60.5 to 31.0]

20. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: Large LDL Particles
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for Large LDL Particles.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nmol/L | 411 (247) | 501 (302)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.0034, ANOVA; Mean Difference (Net) = -135.3, 95% CI 2-sided [-224.7 to -45.8]

21. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12:Total Very Low-Density Lipoprotein (VLDL) and Chylomicron Particles
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for VLDL and Chylomicron Particles.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nmol/L | 24.8 (18.5) | 37.3 (24.7)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.0129, ANOVA; Mean Difference (Net) = -10.0, 95% CI 2-sided [-17.9 to -2.2]

22. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: Total HDL Particles
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for Total HDL Particles.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: micromol/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
micromol/L | 29.79 (4.699) | 30.92 (5.940)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.3088, ANOVA; Mean Difference (Net) = -0.77, 95% CI 2-sided [-2.26 to 0.72]

23. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: LDL Particle Size
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for LDL Particle size.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nm
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nm | 20.94 (0.546) | 20.89 (0.549)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.6905, ANOVA; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.15 to 0.23]

24. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: VLDL Particle Size
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for VLDL Particle Size.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nm
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 67 | 34
nm | 52.27 (7.063) | 51.33 (8.801)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.5008, ANOVA; Mean Difference (Net) = 0.96, 95% CI 2-sided [-1.86 to 3.78]

25. Secondary Outcome: Mean Change in Lipid Particle Concentration From Baseline To Week 12: HDL Particle Size
Description: The effect of once-daily oral dosing of MGL-3196 versus placebo for 12 weeks in terms of change from baseline was assessed for HDL Particle Size.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: nm
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 35
nm | 9.30 (0.589) | 9.19 (0.586)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; Test type: Superiority; p = 0.1066, ANOVA; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.03 to 0.26]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 12
Arm/Group | MGL-3196 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/78 | 1/38
Other Adverse Events (participants affected / at risk) | 65/78 | 28/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MGL-3196 (N=78) | Placebo (N=38)
Pyrexia (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MGL-3196 (N=78) | Placebo (N=38)
Diarrhea (Gastrointestinal disorders) | 15 | 4
Nausea (Gastrointestinal disorders) | 16 | 2
Abdominal Pain (Gastrointestinal disorders) | 5 | 2
Flatulence (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 8 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 0
Hepatic enzyme increased (Investigations) | 7 | 0
Nasopharyngitis (Infections and infestations) | 10 | 6
Headache (Nervous system disorders) | 10 | 6
Dizziness (Nervous system disorders) | 4 | 4
Fatigue (General disorders) | 7 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release up to 45 days prior to submission and can embargo communications regarding study results for a period that is more than 90 days from the date that the communication is submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT03038022/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT03038022/SAP_001.pdf